CLINICAL TRIAL: NCT00818896
Title: A Model Statewide Trial to Detect and Treat Maternal Hypothyroidism in Pregnancy
Brief Title: Maternal Hypothyroidism in Pregnancy
Status: Completed | Type: Observational
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, James Haddow, MD, Dr. James Haddow, Women and Infants Hospital of Rhode Island
Other Study IDs: IRB #08-0005; R18DP001148 (NIH)
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Hypothyroidism
Keywords: thyroid deficiency; pregnancy; post-partum thyroid dysfunction; permanent hypothyroidism
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and urine samples from women who consent are to be stored in the freezer. Iodine measurements will be performed in urine samples and, possibly, serum samples. Consent is also asked for use of stored samples for other research purposes in the future.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There is general agreement that thyroid gland function should be assessed in pregnant women. When the gland produces too little thyroid hormone (hypothyroidism), all of the woman's bodily functions slow down, and there are problems with her baby's development. Until now, physicians have identified this problem on an individual basis (case-finding), but this approach misses many of the cases. Our trial aims to replace case-finding with a routine blood test that is highly effective at detecting hypothyroidism, thereby allowing treatment to correct the deficiency. This approach can eventually be implemented throughout the United States.

DETAILED DESCRIPTION:
This is a model community-based trial in Rhode Island (RI), aimed at avoiding or minimizing morbidity from overt maternal hypothyroidism by systematic detection and treatment, beginning at the 1st prenatal visit. This model can be superimposed on existing prenatal screening programs and is intended ultimately to replace "case-finding", which has recently been shown ineffective. Three aspects of maternal and child health are compromised when a pregnant woman is thyroid deficient: 1) the woman's own health and well-being; 2) her baby's brain development; and 3) overall health of the pregnancy (e.g., fetal death, prematurity, preeclampsia). Thyroid stimulating hormone (TSH) measurement, a well accepted indicator of thyroid dysfunction, will serve as the primary test for both diagnosis and monitoring. A TSH value >10 mU/L indicates overt hypothyroidism. Among the state's 14,000 annual pregnancies, 42 women (0.3%) will be overtly hypothyroid early in gestation (32 undiagnosed, and 10 under-treated). TSH values between 4.5 mU/L (98th centile) and 9.9 mU/L indicate subclinical hypothyroidism. The 240 women in this category will also receive treatment, and information will be gathered about disease progression to inform future practice. Approximately half of all RI's pregnancies are cared for by practices in Greater Providence, and TSH testing will initially be introduced, there. The research component is also within that area. Testing will subsequently be extended to the entire state. The program is centrally managed by three units at Women and Infants Hospital, in consultation with RI's Birth Defects Program Director. Program goals are to: provide TSH testing to at least 70% of pregnant women in Greater Providence; provide TSH testing to at least 50% of pregnant women elsewhere in RI; test 70% of screened women by 12 weeks' gestation, and 90% by 18 weeks' gestation; begin treatment in Greater Providence by 13 weeks' in 70%, and by 19 weeks' in 90%; document successful treatment during pregnancy in 90% (TSH >0.1 mU/L and <2.0 mU/L; retain 95% treated women to end of pregnancy, and 90% for up to 1 year postpartum; obtain pregnancy complications and birth outcomes for the entire cohort (Vital Records).

Data will be collected on participation by practices and women, % of women with undiagnosed thyroid deficiency, compliance with follow-up and treatment during pregnancy and for up to one year afterwards, outcomes of their pregnancies, % of hypothyroid women with postpartum thyroid dysfunction, % of women with subclinical hypothyroidism who remain hypothyroid one year postpartum, physician attitudes, and program costs.

ELIGIBILITY:
Inclusion Criteria:

* TSH value >98th centile in early pregnancy

Exclusion Criteria:

* Women with known hypothyroidism

Ages: 17 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The subjects will be 176 pregnant women and adolescents discovered to have varying degrees of hypothyroidism during the first and early second trimesters. This disorder will be identified by a blood test offered as part of routine prenatal care in a CDC-sponsored community-based program at prenatal practices in Providence, Rhode Island. These 176 women all will receive appropriate treatment for their hypothyroidism, and permission will be sought to record information about the natural history of their condition during the first postpartum year, as a way to inform future practice. The women will range in age from about 17 to 44 years. Their racial/ethnic composition will reflect that of the general population of Rhode Island.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2008-04; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Percent of women who develop permanent hypothyroidism. | Up to two years

SECONDARY OUTCOMES:
Percent of women with post-partum thyroid dysfunction. | Up to two years

CONTACTS AND LOCATIONS:
Overall Officials: James E. Haddow, M.D., Principal Investigator — Women & Infants Hospital
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States